CLINICAL TRIAL: NCT05410743
Title: A Phase 1/2, Non-Randomized, Open-Label, Dose Escalation, Single-Center Study to Determine the Safety, Bio-distribution, and Preliminary Effectiveness and Efficacy of 177Lu-TATE-EB-01（LNC1010）in Adult Subjects with SSTR2-positive Tumors
Brief Title: Evaluation of 177Lu-TATE-EB-01（LNC1010）in SSTR2-positive Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022KY051
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-09

CONDITIONS: SSTR2-positive Tumors
Keywords: SSTR2-positive tumors; 177Lu; LNC1010; SSTR antagonist

STUDY DESIGN:
Intervention Model Description: phase 1 To evaluate response to the different groups with doses of 2.22 GBq(60 mCi) and 3.33GBq (90 mCi) and 4.99 GBq (135mCi) of 177Lu-LNC1010 in patients with advanced or metastatic SSTR2-positive tumors;Phase 2 will reassess treatment efficacy and safety using a fixed dose identified in Phase 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 177Lu-LNC1010 1 (Experimental): The patients were intravenously injected with single dose 2.22GBq (60 mCi) of 177Lu-LNC1010 and underwent 68Ga-DOTA-TATE PET/CT scans before and after the treatment.
  Interventions: Drug: 177Lu-LNC1010 1
- 177Lu-LNC1010 2 (Experimental): The patients were intravenously injected with single dose 3.33GBq (90 mCi) of 177Lu-LNC1010 and underwent 68Ga-DOTA-TATE PET/CT scans before and after the treatment.
  Interventions: Drug: 177Lu-LNC1010 2
- 177Lu-LNC1010 3 (Experimental): The patients were intravenously injected with single dose 4.99 GBq (135mCi) of 177Lu-LNC1010 and underwent 68Ga-DOTA-TATE PET/CT scans before and after the treatment.
  Interventions: Drug: 177Lu-LNC1010 3
- 177Lu-LNC1010 4 (Experimental): Patients received a single, fixed dose of 177Lu-LNC1010 via intravenous injection, utilizing the well-tolerated and safe dose identified in Phase 1. They also underwent 68Ga-DOTA-TATE PET/CT scans both before and after the treatment to monitor their response.
  Interventions: Drug: 177Lu-LNC1010 4

INTERVENTIONS:
Drug: 177Lu-LNC1010 1 — The patients were intravenously injected with single dose 2.22GBq (60 mCi) of 177Lu-LNC1010 and underwent 68Ga-DOTA-TATE PET/CT scans before and after the treatment.
  Arms: 177Lu-LNC1010 1
Drug: 177Lu-LNC1010 2 — The patients were intravenously injected with single dose 3.33GBq （90 mCi) of 177Lu-LNC1010 and underwent 68Ga-DOTA-TATE PET/CT scans before and after the treatment.
  Arms: 177Lu-LNC1010 2
Drug: 177Lu-LNC1010 3 — The patients were intravenously injected with single dose 4.99GBq (135 mCi) of 177Lu-LNC1010 and underwent 68Ga-DOTA-TATE PET/CT scans before and after the treatment.
  Arms: 177Lu-LNC1010 3
Drug: 177Lu-LNC1010 4 — Patients received a single, fixed dose of 177Lu-LNC1010 via intravenous injection, utilizing the well-tolerated and safe dose identified in Phase 1. They also underwent 68Ga-DOTA-TATE PET/CT scans both before and after the treatment to monitor their response.
  Arms: 177Lu-LNC1010 4

SUMMARY:
177Lu-LNC1010(177Lu-EB-TATE-01) is a radiotherapeutic drug indicated in subjects with unresectable, metastatic somatostatin receptor (SSTR) positive tumors.

In this study, we designed and developed a new radioligand, EB-TATE-01 (second generation long-acting EB-TATE formula), through combining EB and altering the linker to further improve the pharmacokinetics and pharmacodynamics, leading to substantially enhanced radioligand therapy effect.

This is an open-label, non-controlled, non-randomized study to investigate the long-lasting radiolabeled somatostatin analogue based peptide receptor radionuclide therapy and evaluate response to 177Lu-LNC1010 in patients with advanced SSTR2-positive tumors. Different groups with doses of 2.22GBq (60 mCi), 3.33GBq (90mCi) and 4.99GBq (145mCi) of 177Lu-LNC1010 will be injected intravenously. All patients will undergo 68Ga-DOTA-Octreotide(TATE) PET/CT scans before and after the treatment.

DETAILED DESCRIPTION:
Somatostatin receptor(SSTR), especially SSTR subtype 2 (SSTR2),has been a popular target for molecular imaging and radionuclide therapy in recent years. SSTR antagonists, such as LNC1010, have emerged as a new type of somatostatin analog, characterized by a low internalization rate and high tumor affinity. 68Ga-DOTA(68Ga-DOTA)-LNC1010 has been reported that it showed favorable biodistribution, high tumor uptake, and good tumor retention, resulting in high image contrast. SSTR2 has been found highly expressed in SSTR2-positive tumors, indicating the feasibility of Positron Emission Tomography（PET)/ CT with 68Ga-DOTA-conjugated peptides for imaging SSTR2 expression and peptide-receptor radionuclide therapy (PRRT) for the treatment option in SSTR2-positive tumors. However, a major problem in the therapeutic use of 177Lu-DOTA(177Lu-DOTA)-LNC1010 has been its short half-life and fast rate of clearance.

This combined phase 1/2 clinical trial is designed to initially investigate the safety, tolerability, pharmacokinetics, dosimetry, and preliminary efficacy of 177Lu-LNC1010 in patients with advanced or metastatic SSTR2-positive tumors during the phase 1 portion. The objective is to establish a well-tolerated dose with acceptable side effects. Following this, the phase 2 portion of the trial will involve repeated administration of 177Lu-LNC1010 PRRT at the identified safe fixed dose, aiming to maximize the treatment effect while ensuring patient safety. This phase is set to rigorously evaluate the therapeutic efficacy and potential toxicity of 177Lu-LNC1010 in the management of advanced or metastatic SSTR2-positive tumors.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Histologically proven or cytologically confirmed SSTR positive cancers;
* Measurable disease as defined by Response Criteria in Solid Tumors (RECIST) version 1.1;
* Overexpression of somatostatin receptors of the target lesions at 68Ga-DOTA-TATE positron emission tomography (PET)/computed tomography (CT) with standard uptake value(SUV) of lesions greater than normal liver in at least 1 lesion;
* Patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* Women who are pregnant or breastfeeding;
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 177Lu-EB-TATE as assessed from medical records;
* Previous radioligand treatment with 177Lu-DOTA-TATE;
* Participant has had prior chemotherapy, targeted cancer therapy, immunotherapy, or treatment with an investigational anticancer agent within 4 weeks or 4 half-lives whichever is longer, before the first administration of study drug;
* Participant has not fully recovered from major surgery or significant traumatic injury prior the first dose of study drug or expects to have major surgery during the study period or within 3 months after the last dose of study drug;
* Life expectancy < 3 months as assessed by the treating physician;
* Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements;
* The inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Phase 1-Incidence of treatment-related adverse events (safety and tolerability) | At the end of Cycle 2 (each cycle is 56 days)
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.Dose-limiting toxicity was defined as any 177Lu-DOTA-EB-FAPI-related AE ≥ grade 3 (G3). For Hemoglobin < 8.0 g/dL; < 4.9 mmol/L; < 80 g/L; Need blood transfusion heal. Severe hypocytosis or with this age group The total number of normal cells was reduced >50% and ≤75%.
Phase 2-Efficacy | At the end of Cycle 4 (each cycle is 56 days)
  Patients received a single, fixed dose of 177Lu-LNC1010 via intravenous injection, utilizing the well-tolerated and safe dose identified in Phase 1.68Ga-DOTATATE will be performed for efficacy evaluation by RECIST 1.1. Particularly, 68Ga-DOTATATE will be performed at baseline, and 8 weeks after two treatment cycles.

SECONDARY OUTCOMES:
Phase-1 Dosimetry | At the end of Cycle 1 (each cycle is 56 days)
  Dosimetry, measured as absorbed dose in tumor and normal organs (Gy/GBq), was estimated in the first treatment cycle for each patient.
Phase 1-Overall response rate (ORR) | At the end of Cycle 2 (each cycle is 56 days)
  68Ga-DOTATATE will be performed for efficacy evaluation by RECIST 1.1. Particularly, 68Ga-DOTATATE will be performed at baseline, and 8 weeks after two treatment cycles.
Phase-2 Progression-free survival | baseline, every 8 weeks up to 1 year after last patient first treatment
  Progression-free survival is defined as the time from the date of first dose to the date of the first documented radiological progression or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu W, Cheng Y, Jia R, Zhao H, Bai C, Xu J, Yao S, Huo L. A Prospective, Randomized, Double-Blind Study to Evaluate the Safety, Biodistribution, and Dosimetry of 68Ga-NODAGA-LM3 and 68Ga-DOTA-LM3 in Patients with Well-Differentiated Neuroendocrine Tumors. J Nucl Med. 2021 Oct;62(10):1398-1405. doi: 10.2967/jnumed.120.253096. Epub 2021 Feb 12. PMID 33579804